CLINICAL TRIAL: NCT04456751
Title: Is a Reintervention for Pediatric Cardiac Surgery Associated With Higher Blood Transfusion Requirements ?
Brief Title: Is Redo Pediatric Cardiac Surgery a Risk Factor for Transfusion?
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Head of Anesthesiology department, Brugmann University Hospital
Other Study IDs: CHUB_redoped
Record Dates: First submitted 2020-06-25; First posted 2020-07-02 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Pediatric Cardiac Surgery; Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No redo op: Patients with a single cardiac operation under extracorporeal bypass
- Redo op: Patients with a redo cardiac operation under extracorporeal bypass
  Interventions: Other: Redo op

INTERVENTIONS:
Other: Redo op — Patients with a redo operation
  Groups: Redo op

SUMMARY:
In pediatric cardiac surgery, transfusion requirements are associated with age, development status, pathology, type of surgical intervention and extracorporeal bypass. In adult cardiac surgery, reinterventions (redo)are clearly linked to higher transfusion rates. The investigators want to study if this association is also true in pediatric cardiac surgery.

DETAILED DESCRIPTION:
Whereas in adult cardiac surgery, redo-interventions are clearly linked to a higher transfusion rate, this is not really known in paediatric cardiac surgery. In this retrospective study, the investigators will analyse our database for paediatric cardiac surgery patients aged 0-16 years and operated between 2002 and 2017. Patients with a single cardiac surgery will be compared to patients with a second cardiac operation under extracorporeal bypass. The investigators will test the variables for normal distribution using a Shapiro-Wilk test. Non normal distributed variables will be compared by a non-parametric test (Mann Whitney U), frequency analysis will be done by a Chi-Square test. A univariate analysis will determine predicting factors for transfusion. Factors with a P value < 0.1 will be analysed by a multivariate analysis to determine independent factors for transfusion. Odds with 95% confidence intervals will be calculated. A P value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 0 and 16 years
* Cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* Jehova's witness

Max Age: 16 Years | Sex: All
Age Groups: Child
Study Population: All patients between 0 and 16 years undergoing cardiac surgery with cardiopulmonary bypass in our institution. We will exclude Jehovah's witness patient as they refuse a transfusion.
Sampling Method: Non-Probability Sample
Enrollment: 2439 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Transfusion of packed red cells (mL/kg) | Day of operation up to 5 days postop
  Transfusion requirements will be measured as volume of packed red cells given as mL packed red cells/kg of body weight

CONTACTS AND LOCATIONS:
Overall Officials: Denis Schmartz, MD, Principal Investigator — CHU Brugmann
Locations (1):
- Hôpital Universitaire des Enfants Reine Fabiola, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No